CLINICAL TRIAL: NCT00804453
Title: Evaluation of the Biocompatibility of Cartridge Blood Set Versus Standard Blood Line: A Pilot Monocentric Open Randomized and Cross-over Study.
Brief Title: Evaluation of the Biocompatibility of Cartridge Blood Set Versus Standard Blood Line
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vantive Health LLC (Industry)
Collaborators: Gambro Lundia AB (Industry); Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1455; ISRCTN15261860
Record Dates: First submitted 2008-12-05; First posted 2008-12-08 (Estimated); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Chronic Kidney Failure
Keywords: Chronic Kidney Failure; Hemodialysis; Biocompatibility
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Standard blood line
  Interventions: Device: Standard blood line
- 2 (Experimental): Cartridge blood line
  Interventions: Device: Cartridge blood set

INTERVENTIONS:
Device: Cartridge blood set — Once a week
  Arms: 2
Device: Standard blood line — Once a week
  Arms: 1

SUMMARY:
The primary objective is to collect data to evaluate the biocompatibility of two types of blood circuit, already on the market.

DETAILED DESCRIPTION:
Interactions between blood components (cells and proteins) and the extracorporeal circuit induce the activation of several biological systems such as platelets, complement and coagulation cascades. The coagulation system generates a key enzyme, factor IIa or thrombin, responsible for blood clotting in the dialysis circuit Because clotting in the circuit may reduce the dialysis efficiency, the anticoagulation of the extracorporeal circuit is needed .

For several years, most of the researches were mainly focused on the improvement of the biocompatibility of dialysis membranes .

The contribution of the various components of the dialysis circuit on the coagulation activation has not been clearly established.

A circuit integrating a cartridge blood set is commercialised for several years. The design of this cartridge blood set reduces the surface in contact with blood and minimizes the blood air interface which are well known sources of coagulation activation.

The aim of this study is to collect data to evaluate the biocompatibility of two types of blood circuit (cartridge blood set vs standard blood line).

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from chronic renal failure,
* Patients treated in HD performed with or without heparin injection in the extra corporeal circuit (ECC) irrespective the type of heparin (UFH and LMWH),
* Patients treated three times a week for a minimum of three (3) months,
* Patients 18 years or older,
* Patients with a well-functioning vascular access as judged by the investigator,
* Patients with negative serologies (HIV, hepatitis),
* Patients having signed written informed consent to participate in the study.

Exclusion Criteria:

* Patients with known allergy to heparin,
* Patients with acute inflammatory event that may affect, as judged by the investigator, the results of the study or the safety of the patients,
* Active malignant disease,
* Pregnant women, nursing mothers and women planning a pregnancy during the course of the study,
* Patients under guardianship,
* Patients participating in other studies that could interfere with the objectives of this study,
* Patients treated in single needle mode,
* Patients with catheter,
* Patients receiving Anti-Vit K drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-11; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
The biocompatibility will be followed, during dialysis treatment, by measuring TAT complex generation. | During dialysis treatment

SECONDARY OUTCOMES:
The quality of the restitution of both the filter and the circuit, at the end of each treatment, will be evaluated via visual scales. | End of dialysis treatment

CONTACTS AND LOCATIONS:
Overall Officials: Walid Arkouche, Dr, Principal Investigator — AURAL dialysis centre Lyon France
Locations (1):
- AURAL, Bourgoin, France

REFERENCES:
- [Background] Lucchi L, Ligabue G, Marietta M, Delnevo A, Malagoli M, Perrone S, Stipo L, Grandi F, Albertazzi A. Activation of coagulation during hemodialysis: effect of blood lines alone and whole extracorporeal circuit. Artif Organs. 2006 Feb;30(2):106-10. doi: 10.1111/j.1525-1594.2006.00188.x. PMID 16433843